CLINICAL TRIAL: NCT01825096
Title: Multi-Modal fMRI/NIRS for Estimation of CMRO2 for Neuroimaging Studies of Drug Abuse and Psychiatric Illness Problems
Brief Title: Simultaneous FMRI and NIRS to Estimate Brain Cerebral Metabolism
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Lisa Nickerson, PhD, Assistant Physicist, Mclean Hospital
Other Study IDs: 2012p00622
Record Dates: First submitted 2013-03-27; First posted 2013-04-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: cerebral metabolism; functional magnetic resonance imaging; near infrared spectroscopy

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- baseline: No intervention. Participants are scanned at baseline.

SUMMARY:
The principal advantages of functional magnetic resonance imaging (fMRI) with blood-oxygenation- level-dependent (BOLD) contrast for studying brain function are: non-invasiveness, ubiquitous availability, relatively high spatiotemporal resolution, and the ability to map function over the entire brain. Thus, BOLD fMRI is the most widely applied technology to study healthy brain function and pathophysiology associated with disease. In studies of drug abuse and psychiatric illness though, normal assumptions mapping BOLD signals to neurometabolism may be violated. Generally, these effects are ignored, resulting in large study-to-study variability.

Quantitative fMRI (qfMRI) measures metabolism directly and is more suitable for studies of drug abuse and psychiatric illness. However, qfMRI is too complex for routine use. Cerebral metabolism during brain activation during visual stimulation measured with a new fMRI approach that is simple enough for clinical applications will be compared to CMRO2 activation measured using standard qfMRI.

DETAILED DESCRIPTION:
Healthy subjects will undergo a single imaging session. During the imaging session, fMRI and simultaneous near-infrared spectroscopy measurements will be made during visual stimulation (e.g., viewing a flashing checkerboard). This is a methods development study focused on comparing a new method for estimating CMRO2 associated with brain activation with the standard fMRI approach for estimating CMRO2.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 to 40 years old
* Physically healthy by self-report

Exclusion Criteria:

Diagnosis of current drug abuse/dependence, including nicotine, as assessed by DSM-IV criteria

* Current diagnosis of Axis I disorder using DSM-IV criteria, or any Axis I disorder within past 5 years
* Current daily use of antipsychotic, antidepressant, or other psychoactive prescription drug, as well as daily use of non-prescription drugs
* Life threatening or unstable medical illness, or one that can create marked change in mental state
* Heavy caffeine use (greater than 300 mg on a regular, daily basis)
* History of seizure disorder
* Subjects that report any history or current major medical illness (cardiovascular, pulmonary, psychiatric, or neurological disorders)
* Subjects who have metal in their body or suffer from claustrophobia cannot participate in this research study.
* Additional MR exclusion criteria may include people with:
* Cardiac pacemakers
* Metal clips on blood vessels (also called stents)
* Artificial heart valves
* Artificial arms, hands, legs, etc.
* Brain stimulator devices
* Implanted drug pumps
* Ear implants
* Eye implants or known metal fragments in eyes
* Exposure to shrapnel or metal filings (wounded in military combat, sheet metal workers, welders, and others)
* Other metallic surgical hardware in vital areas
* Certain tattoos with metallic ink (subjects are asked to inform research staff if they have a tattoo)
* Metal Containing Intrauterine Devices (IUDs).
* Certain transdermal (skin) patches such as Transderm Scop (scopolamine for motion sickness).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1 healthy subject will be recruited for the study from the general population to undergo 12 separate study visits.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in brain activity associated with visual stimulation | cross-sectional, start and up to 6 minutes
  CMRO2 brain activation in visual cortex associated with visual stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Nickerson, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Imaging Center, Belmont, Massachusetts, United States